CLINICAL TRIAL: NCT06093763
Title: Evaluating the Utility of Bone Grafts in Open Wedge Corrective Osteotomy and Plate Fixation in Patients With Malunited Distal Radius Fractures
Brief Title: Evaluating the Utility of Bone Grafts in Open Wedge Corrective Osteotomy and Plate Fixation
Acronym: WOPPeR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Haga Hospital (Other); Amsterdam UMC (Other); VieCuri Medical Centre (Other); Zuyderland Medical Centre (Other); Elkerliek Hospital (Other); Erasmus Medical Center (Other); Amphia Hospital (Other); Reinier Haga Orthopedisch Centrum (Other); Flevoziekenhuis (Other); Diakonessenhuis, Utrecht (Other); Xpert Clinics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL68126.068.18
Record Dates: First submitted 2023-10-10; First posted 2023-10-23 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2023-10

CONDITIONS: Malunion of Fracture of Radius
Keywords: open wedge osteotomy; bone grafting; time of bone healing; complications; Quality of life; Subjective and objective functional outcomes; Cost effectiveness
MeSH Terms: interventions — Population Groups; Bone Transplantation

STUDY DESIGN:
Intervention Model Description: All included patients will undergo an open wedge osteotomy and plate fixation according to the standard surgical techniques. In one group, the bone defect will be filled with bone graft of the iliac crest after open wedge osteotomy according the standard procedure. The other group includes patients who will not receive any bone grafts. The participating hospitals have extensive experience with both treatments.
Who Masked: Participant
Masking Description: A web based randomisation tool will used for randomization according to the GCP-guidelines. Prestratification per hospital will be performed. Patients and the treating surgeon cannot be blinded for the treatment because a part of these patients will undergo bone grafting derived from the iliac crest. The statistician will be blinded for the treatment.
  6.3 Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with symptomatic malunion of distal radius receiving bone grafting (Active Comparator): Open wedge corrective osteotomy and plate fixation with harvesting and using bone from the iliac crest.
  Interventions: Procedure: Group with bone grafting
- Patients with symptomatic malunion of distal radius receiving none bone grafts (Active Comparator): Open wedge corrective osteotomy and plate fixation without harvesting and using bone from the iliac crest.
  Interventions: Procedure: Group without bone grafting

INTERVENTIONS:
Procedure: Group without bone grafting — Open wedge corrective osteotomy and plate fixation without bone grafting.
  Arms: Patients with symptomatic malunion of distal radius receiving none bone grafts
Procedure: Group with bone grafting — Open wedge corrective osteotomy and plate fixation with harvesting and using bone from the iliac crest.
  Arms: Patients with symptomatic malunion of distal radius receiving bone grafting

SUMMARY:
INTRODUCTION A variety of bone grafts and substitutes are available for filling bone defects in the distal radius after corrective osteotomy, but the harvesting of bone from the iliac crest is the gold standard as it allows easy access to corticocancellous bone of a desirable quality and quantity. The idea behind bone grafting is to provide optimal bone formation and structural stability, which is crucial for bone healing. However, the harvesting and use of bone from the iliac crest potentially comes with the risk of complications such as delayed union of the osteotomy defect; size mismatch between the graft and the osteotomy defect; longer operation time; donor site morbidity including nerve, arterial, and ureteral injury; herniation of abdominal contents; sacroiliac joint instability; pelvic fractures; hematoma and infection. As these disadvantages of bone grafting can have a major impact on patients' everyday lives, research is needed on whether bone grafting is genuinely necessary during corrective osteotomy and plate fixation of the distal radius

OBJECTIVE The objective of this study is to investigate whether harvested bone graft from the iliac crest necessary is during corrective osteotomy and plate fixation in patients with malunited distal radius fractures.

STUDY DESIGN This is a prospective, randomized, controlled multicenter study. Patients will undergo the following examinations once before the operation and five times afterwards: 1) the patients will fill out three questionnaires, 2) complications will be noted, 3) the wrist function will be measured, and 4) radiographs/CT scans will be made.

STUDY POPULATION All patients over the age of 18 years who have a symptomatic malunion after distal radius fracture and are eligible for surgical correction.

INTERVENTION Surgical correction in the form of open wedge corrective osteotomy and plate fixation without bone grafting.

USUAL CARE Open wedge corrective osteotomy and plate fixation with harvesting bone from the iliac crest.

OUTCOME MEASURES Primary outcomes: complications and quality of life. Secondary outcomes: time to complete bone healing, functional outcomes, and cost effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex over the age of 18 years
* Symptomatic malunion of the distal radius
* Eligible for open wedge osteotomy and plate fixation with or without bone grafting from iliac crest.
* Patients are able to undergo postoperative follow-up of at least 12 months.

Exclusion Criteria:

* Patients who are pregnant
* Patients who have known systemic or metabolic disorders leading to progressive bone deterioration
* Patients who take chronic use of glucocorticoids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Complications | follow-up period of at least one year
  number and severity during and after the operation
Quality of life using the EQ-5D-5L questionnaire | follow-up period of one year
  EQ-5D-5L questionnaire
Time to complete bone healing | follow-up period of one year
  Bone healing will be considered complete when the osteotomy gap is filled with bone formation.

SECONDARY OUTCOMES:
Subjective functional outcomes | follow-up period of one year
  Disability of the Arm, Shoulder and Hand Questionnaire (DASH): measure of self-rated upper-extremity disability and symptoms in activities of daily living
Subjective functional outcome | follow-up period of one year
  Patient-Rated Wrist Evaluation (PRWE) Questionnaire: measure of self-rated wrist pain and disability in activities of daily living
Objective functional outcomes | follow-up period of one year
  Active range of motion
Cost effectiveness | follow-up period of at least one year
  cost-effectiveness analysis

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Hannemann, MD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- MaastrichtUMC, Maastricht, Zuid-Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No